CLINICAL TRIAL: NCT00960440
Title: Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Of The Safety And Efficacy Of 2 Doses Of CP-690,550 In Patients With Active Rheumatoid Arthritis On Background Methotrexate With Inadequate Response To TNF Inhibitors
Brief Title: Study of CP-690,550 Versus Placebo In Rheumatoid Arthritis Patients On Background Methotrexate With Inadequate Response To Tumor Necrosis Factor (TNF) Inhibitors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921032
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Results first posted 2013-01-10 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Arthritis, Rheumatoid
Keywords: randomized double-blind placebo-controlled investigational drug oral therapy safety and efficacy
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib; Double-Blind Method

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sequence 1 (Experimental)
  Interventions: Drug: CP-690,550
- Sequence 2 (Experimental)
  Interventions: Drug: CP-690,550
- Sequence 3 (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: CP-690,550
- Sequence 4 (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: CP-690,550

INTERVENTIONS:
Drug: CP-690,550 — Oral tablets administered at 5 mg BID daily for 6 months during the double-blind, placebo-controlled period.
  Arms: Sequence 1
Drug: CP-690,550 — Oral tablets administered at 10 mg BID daily for 6 months during the double-blind, placebo-controlled period.
  Arms: Sequence 2
Drug: Placebo — Oral placebo tablets administered BID daily during the first 3 months of the double-blind, study period.
  Other Names: double-blind, placebo-controlled phase
  Arms: Sequence 3
Drug: CP-690,550 — Oral tablets administered at 5 mg BID daily during the second 3 months of the double-blind, study period.
  Other Names: double-blind, extension phase
  Arms: Sequence 3
Drug: Placebo — Oral placebo tablets administered BID daily during the first 3 months of the double-blind, placebo-controlled period.
  Other Names: double-blind, placebo-controlled phase
  Arms: Sequence 4
Drug: CP-690,550 — Oral tablets administered at 10 mg BID daily during the second 3 months of the double-blind, study period.
  Other Names: double-blind, extension phase
  Arms: Sequence 4

SUMMARY:
This study will test if CP-690,550 is safe and effective in rheumatoid arthritis patients taking methotrexate who have an inadequate response to tumor necrosis factor inhibitor treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults with moderate to severe rheumatoid arthritis on a stable dose of methotrexate who have inadequate response to Tumor Necrosis Factor (TNF) inhibitors.

Exclusion Criteria:

* Pregnancy, severe acute or chronic medical conditions, including serious infections or clinically significant laboratory abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2009-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (81):
- United States (32):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Farmington, Connecticut
  - Pfizer Investigational Site, Trumbull, Connecticut
  - Pfizer Investigational Site, Aventura, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Boise, Idaho
  - Pfizer Investigational Site, Idaho Falls, Idaho
  - Pfizer Investigational Site, Springfield, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Portland, Maine
  - Pfizer Investigational Site, Cumberland, Maryland
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Flowood, Mississippi
  - Pfizer Investigational Site, Tupelo, Mississippi
  - Pfizer Investigational Site, Lebanon, New Hampshire
  - Pfizer Investigational Site, Voorhees Township, New Jersey
  - Pfizer Investigational Site, Rocky Mount, North Carolina
  - Pfizer Investigational Site, Bethlehem, Pennsylvania
  - Pfizer Investigational Site, Willow Grove, Pennsylvania
  - Pfizer Investigational Site, Wyomissing, Pennsylvania
  - Pfizer Investigational Site, Hixson, Tennessee
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Lubbock, Texas
  - Pfizer Investigational Site, Vancouver, Washington
- Australia (3):
  - Pfizer Investigational Site, Kogarah, New South Wales
  - Pfizer Investigational Site, Daw Park, South Australia
  - Pfizer Investigational Site, Heidelberg, Victoria
- Pfizer Investigational Site, Vienna, Austria
- Belgium (4):
  - Pfizer Investigational Site, Genk
  - Pfizer Investigational Site, Hasselt
  - Pfizer Investigational Site, Kortrijk
  - Pfizer Investigational Site, Liège
- Brazil (4):
  - Pfizer Investigational Site, Goiânia, Goiás
  - Pfizer Investigational Site, Curitiba, Paraná
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo, São Paulo
- Canada (5):
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Pointe-Claire, Quebec
- France (4):
  - Pfizer Investigational Site, Amiens
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Orléans
  - Pfizer Investigational Site, Paris
- Germany (9):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Cologne
  - Pfizer Investigational Site, Erlangen
  - Pfizer Investigational Site, Frankfurt am Main
  - Pfizer Investigational Site, Halle
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Rheine
  - Pfizer Investigational Site, Würzburg
- Ireland (2):
  - Pfizer Investigational Site, Croom, Co. Limerick
  - Pfizer Investigational Site, Dublin
- Italy (2):
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Iesi
- Pfizer Investigational Site, San Juan, Puerto Rico
- South Korea (3):
  - Pfizer Investigational Site, Busan
  - Pfizer Investigational Site, Daegu
  - Pfizer Investigational Site, Seoul
- Spain (7):
  - Pfizer Investigational Site, Santiago de Compostela, A Coruña
  - Pfizer Investigational Site, Mérida, Badajoz
  - Pfizer Investigational Site, Bilbao, Bizkaia
  - Pfizer Investigational Site, Santander, Cantabria
  - Pfizer Investigational Site, Barakaldo, Vizcaya
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Valencia
- Taiwan (4):
  - Pfizer Investigational Site, Niao Sung Hsiang, Kaohsiung County
  - Pfizer Investigational Site, Kweishan, Taoyuan County
  - Pfizer Investigational Site, Changhua
  - Pfizer Investigational Site, Kaohsiung City

REFERENCES:
- [Derived] Hetland ML, Strangfeld A, Bonfanti G, Soudis D, Deuring JJ, Edwards RA. Machine learning prediction and explanatory models of serious infections in patients with rheumatoid arthritis treated with tofacitinib. Arthritis Res Ther. 2024 Aug 27;26(1):153. doi: 10.1186/s13075-024-03376-9. PMID 39192350
- [Derived] Wright GC, Mysler E, Kwok K, Cadatal MJ, Germino R, Yndestad A, Kinch CD, Ogdie A. Impact of Race on the Efficacy and Safety of Tofacitinib in Rheumatoid Arthritis: Post Hoc Analysis of Pooled Clinical Trials. Rheumatol Ther. 2024 Oct;11(5):1135-1164. doi: 10.1007/s40744-024-00677-y. Epub 2024 Jul 3. PMID 38958913
- [Derived] Citera G, Jain R, Irazoque F, Madariaga H, Gruben D, Wang L, Stockert L, Santana K, Ebrahim A, Ponce de Leon D. Tofacitinib Efficacy in Patients with Rheumatoid Arthritis and Probable Depression/Anxiety: Post Hoc Analysis of Phase 3 and 3b/4 Randomized Controlled Trials. Rheumatol Ther. 2024 Feb;11(1):35-50. doi: 10.1007/s40744-023-00612-7. Epub 2023 Nov 5. PMID 37925660
- [Derived] Charles-Schoeman C, Hyde C, Guan S, Parikh N, Wang J, Shahbazian A, Stockert L, Andrews J. Relationship Between Paraoxonase-1 Genotype and Activity, and Major Adverse Cardiovascular Events and Malignancies in Patients With Rheumatoid Arthritis Receiving Tofacitinib. J Rheumatol. 2023 Jul 15:jrheum.2023-0112. doi: 10.3899/jrheum.2023-0112. Online ahead of print. PMID 37453736
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Dougados M, Taylor PC, Bingham CO 3rd, Fallon L, Brault Y, Roychoudhury S, Wang L, Kessouri M. The effect of tofacitinib on residual pain in patients with rheumatoid arthritis and psoriatic arthritis. RMD Open. 2022 Sep;8(2):e002478. doi: 10.1136/rmdopen-2022-002478. PMID 36814062
- [Derived] Hansen KE, Mortezavi M, Nagy E, Wang C, Connell CA, Radi Z, Litman HJ, Adami G, Rossini M. Fracture in clinical studies of tofacitinib in rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2022 Dec 27;14:1759720X221142346. doi: 10.1177/1759720X221142346. eCollection 2022. PMID 36601090
- [Derived] Curtis JR, Yamaoka K, Chen YH, Bhatt DL, Gunay LM, Sugiyama N, Connell CA, Wang C, Wu J, Menon S, Vranic I, Gomez-Reino JJ. Malignancy risk with tofacitinib versus TNF inhibitors in rheumatoid arthritis: results from the open-label, randomised controlled ORAL Surveillance trial. Ann Rheum Dis. 2023 Mar;82(3):331-343. doi: 10.1136/ard-2022-222543. Epub 2022 Dec 5. PMID 36600185
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Dikranian AH, Gonzalez-Gay MA, Wellborne F, Alvaro-Gracia JM, Takiya L, Stockert L, Paulissen J, Shi H, Tatulych S, Curtis JR. Efficacy of tofacitinib in patients with rheumatoid arthritis stratified by baseline body mass index: an analysis of pooled data from phase 3 studies. RMD Open. 2022 May;8(1):e002103. doi: 10.1136/rmdopen-2021-002103. PMID 35577477
- [Derived] Dikranian A, Gold D, Bessette L, Nash P, Azevedo VF, Wang L, Woolcott J, Shapiro AB, Szumski A, Fleishaker D, Wollenhaupt J. Frequency and Duration of Early Non-serious Adverse Events in Patients with Rheumatoid Arthritis and Psoriatic Arthritis Treated with Tofacitinib. Rheumatol Ther. 2022 Apr;9(2):411-433. doi: 10.1007/s40744-021-00405-w. Epub 2021 Dec 17. PMID 34921355
- [Derived] Winthrop KL, Curtis JR, Yamaoka K, Lee EB, Hirose T, Rivas JL, Kwok K, Burmester GR. Clinical Management of Herpes Zoster in Patients With Rheumatoid Arthritis or Psoriatic Arthritis Receiving Tofacitinib Treatment. Rheumatol Ther. 2022 Feb;9(1):243-263. doi: 10.1007/s40744-021-00390-0. Epub 2021 Dec 6. PMID 34870800
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Wang L, Chen C, Kwok K, Biswas P, Shapiro A, Madsen A, Wollenhaupt J. Long-term safety of tofacitinib up to 9.5 years: a comprehensive integrated analysis of the rheumatoid arthritis clinical development programme. RMD Open. 2020 Oct;6(3):e001395. doi: 10.1136/rmdopen-2020-001395. PMID 33127856
- [Derived] Strand V, Kaine J, Alten R, Wallenstein G, Diehl A, Shi H, Germino R, Murray CW. Associations between Patient Global Assessment scores and pain, physical function, and fatigue in rheumatoid arthritis: a post hoc analysis of data from phase 3 trials of tofacitinib. Arthritis Res Ther. 2020 Oct 15;22(1):243. doi: 10.1186/s13075-020-02324-7. PMID 33059710
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Kivitz AJ, Cohen S, Keystone E, van Vollenhoven RF, Haraoui B, Kaine J, Fan H, Connell CA, Bananis E, Takiya L, Fleischmann R. A pooled analysis of the safety of tofacitinib as monotherapy or in combination with background conventional synthetic disease-modifying antirheumatic drugs in a Phase 3 rheumatoid arthritis population. Semin Arthritis Rheum. 2018 Dec;48(3):406-415. doi: 10.1016/j.semarthrit.2018.07.006. Epub 2018 Jul 19. PMID 30177460
- [Derived] Hall S, Nash P, Rischmueller M, Bossingham D, Bird P, Cook N, Witcombe D, Soma K, Kwok K, Thirunavukkarasu K. Tofacitinib, an Oral Janus Kinase Inhibitor: Pooled Efficacy and Safety Analyses in an Australian Rheumatoid Arthritis Population. Rheumatol Ther. 2018 Dec;5(2):383-401. doi: 10.1007/s40744-018-0118-2. Epub 2018 Jun 11. PMID 29949132
- [Derived] Mariette X, Chen C, Biswas P, Kwok K, Boy MG. Lymphoma in the Tofacitinib Rheumatoid Arthritis Clinical Development Program. Arthritis Care Res (Hoboken). 2018 May;70(5):685-694. doi: 10.1002/acr.23421. Epub 2018 Apr 2. PMID 28941219
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Thirunavukkarasu K, DeMasi R, Geier J, Kwok K, Wang L, Riese R, Wollenhaupt J. Long-term safety of tofacitinib for the treatment of rheumatoid arthritis up to 8.5 years: integrated analysis of data from the global clinical trials. Ann Rheum Dis. 2017 Jul;76(7):1253-1262. doi: 10.1136/annrheumdis-2016-210457. Epub 2017 Jan 31. PMID 28143815
- [Derived] Vieira MC, Zwillich SH, Jansen JP, Smiechowski B, Spurden D, Wallenstein GV. Tofacitinib Versus Biologic Treatments in Patients With Active Rheumatoid Arthritis Who Have Had an Inadequate Response to Tumor Necrosis Factor Inhibitors: Results From a Network Meta-analysis. Clin Ther. 2016 Dec;38(12):2628-2641.e5. doi: 10.1016/j.clinthera.2016.11.004. Epub 2016 Nov 24. PMID 27889300
- [Derived] Charles-Schoeman C, Burmester G, Nash P, Zerbini CA, Soma K, Kwok K, Hendrikx T, Bananis E, Fleischmann R. Efficacy and safety of tofacitinib following inadequate response to conventional synthetic or biological disease-modifying antirheumatic drugs. Ann Rheum Dis. 2016 Jul;75(7):1293-301. doi: 10.1136/annrheumdis-2014-207178. Epub 2015 Aug 14. PMID 26275429
- [Derived] Strand V, Burmester GR, Zerbini CA, Mebus CA, Zwillich SH, Gruben D, Wallenstein GV. Tofacitinib with methotrexate in third-line treatment of patients with active rheumatoid arthritis: patient-reported outcomes from a phase III trial. Arthritis Care Res (Hoboken). 2015 Apr;67(4):475-83. doi: 10.1002/acr.22453. PMID 25186034
- [Derived] Cohen S, Radominski SC, Gomez-Reino JJ, Wang L, Krishnaswami S, Wood SP, Soma K, Nduaka CI, Kwok K, Valdez H, Benda B, Riese R. Analysis of infections and all-cause mortality in phase II, phase III, and long-term extension studies of tofacitinib in patients with rheumatoid arthritis. Arthritis Rheumatol. 2014 Nov;66(11):2924-37. doi: 10.1002/art.38779. PMID 25047021
- [Derived] Burmester GR, Blanco R, Charles-Schoeman C, Wollenhaupt J, Zerbini C, Benda B, Gruben D, Wallenstein G, Krishnaswami S, Zwillich SH, Koncz T, Soma K, Bradley J, Mebus C; ORAL Step investigators. Tofacitinib (CP-690,550) in combination with methotrexate in patients with active rheumatoid arthritis with an inadequate response to tumour necrosis factor inhibitors: a randomised phase 3 trial. Lancet. 2013 Feb 9;381(9865):451-60. doi: 10.1016/S0140-6736(12)61424-X. Epub 2013 Jan 5. PMID 23294500
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921032&StudyName=Phase%203%2C%20Randomized%2C%20Double-Blind%2C%20Placebo-Controlled%20Study%20Of%20The%20Safety%20And%20Efficacy%20Of%202%20Doses%20Of%20CP-690%2C550%20In%20Patients%20With%20Active%20Rheumatoid%20Arthritis%20On%20Background%20Methotrexate%20With%20Inadequate%20Response%20To%20TNF%20Inhibitors

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-690,550 5 mg: CP-690,550 5 milligram (mg) tablet orally twice daily up to Month 6.
- CP-690,550 10 mg: CP-690,550 10 mg tablet orally twice daily up to Month 6.
- Placebo, Then CP-690,550 5 mg: Placebo matched to CP-690,550 tablet orally twice daily up to Month 3 followed by CP-690,550 5 mg tablet orally twice daily up to Month 6.
- Placebo, Then CP-690,550 10 mg: Placebo matched to CP-690,550 tablet orally twice daily up to Month 3 followed by CP-690,550 10 mg tablet twice daily orally up to Month 6.
Period: Overall Study
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Started | 133 | 134 | 66 | 66
Completed | 107 | 103 | 53 | 48
Not Completed | 26 | 31 | 13 | 18
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Adverse Event | 12 | 12 | 4 | 4
Not completed — Lack of Efficacy | 2 | 5 | 3 | 8
Not completed — Protocol Violation | 2 | 8 | 3 | 4
Not completed — Withdrawal by Subject | 9 | 5 | 2 | 1
Not completed — Other | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- CP-690,550 5 mg: CP-690,550 5 mg tablet orally twice daily up to Month 6.
- Total: Total of all reporting groups
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg | Total
Number analyzed (Participants) | 133 | 134 | 66 | 66 | 399
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (11.5) | 55.1 (11.3) | 54.3 (11.7) | 54.5 (11.0) | 55.0 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 116 | 53 | 53 | 335
  Male | 20 | 18 | 13 | 13 | 64

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Month 3
Description: ACR20 response: greater than or equal to (>=) 20 percent (%) improvement in tender joints count (TJC); >= 20% improvement in swollen joints count (SJC); and >= 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP). For comparison of CP-690,550 with placebo, placebo sequences were combined into single reporting group for Month 3 analysis.
Time Frame: Month 3
Population: Full Analysis Set(FAS):all randomized participants who received at least 1 dose of study treatment, had at least 1 post-baseline measurement. Missing values due to participant dropping due to any reason were imputed using Non-Responder Imputation(NRI). 'N' (Number of Participants Analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Placebo matched to CP-690,550 tablet orally twice daily up to Month 3 followed by CP-690,550 5mg or 10 mg tablet orally twice daily up to Month 6.
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 132 | 133 | 131
percentage of participants | 41.67 | 48.12 | 24.43
Statistical Analysis 1: Comparison: CP-690,550 10 mg vs Placebo; Normal approximation for the difference in binomial proportions was used to test the superiority of CP-690,550 10 mg to placebo and 2-sided 95% confidence interval (CI) was evaluated for the difference in percentages; Test type: Superiority or Other; p < 0.0001, Normal Approximation — A step-down procedure was used to control for multiple comparisons. In order for the comparison to 5 mg to be statistically significant, the comparison to 10 mg had to be statistically significant; Percentage Difference = 23.69, 95% CI 2-sided [12.45 to 34.92], Standard Error of Mean 5.73
Statistical Analysis 2: Comparison: CP-690,550 5 mg vs Placebo; Normal approximation for the difference in binomial proportions was used to test the superiority of CP-690,550 5 mg to placebo and 2-sided 95% CI was evaluated for the difference in percentages; Test type: Superiority or Other; p = 0.0024, Normal Approximation — [p-value comment as in outcome 1, analysis 1]; Percentage Difference = 17.23, 95% CI 2-sided [6.06 to 28.41], Standard Error of Mean 5.70

2. Primary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Month 3
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities:dress/groom;arise;eat; walk;reach;grip; hygiene;common activities over past week. Each item scored on 4-point scale from 0-3:0=no difficulty;1=some difficulty;2=much difficulty;3=unable to do. Overall score was computed as sum of domain scores and divided by number of domains answered. Total possible score range 0-3:0=least difficulty and 3=extreme difficulty. For comparison of CP-690,550 with placebo, placebo sequences were combined into single reporting group for Month 3 analysis.
Time Frame: Baseline, Month 3
Population: FAS included all randomized participants who received at least 1 dose of study treatment and had at least 1 post-baseline measurement. Here 'N' (Number of Participants Analyzed) signifies participants who were evaluable for this measure and 'n' signifies participants who were evaluable at specified time points for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 132 | 134 | 132
Units on a scale
  Baseline (n=132,134,132) | 1.60 (0.66) | 1.50 (0.61) | 1.63 (0.66)
  Change at Month 3 (n=117,125,118) | -0.41 (0.52) | -0.41 (0.52) | -0.17 (0.41)
Statistical Analysis 1: Comparison: CP-690,550 10 mg vs Placebo; Least squares mean difference (LS Mean Difference) and corresponding 95% CI was calculated using a mixed effect repeated measure model with treatment, visit, treatment by visit interaction, and geographic region as fixed effects and participants as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — A step-down procedure was used to control for multiple comparisons. For the comparison of 10 mg to placebo to be statistically significant in this measure, the comparison of 10 mg to placebo in ACR20 had to be significant; LS Mean Difference = -0.28, 95% CI 2-sided [-0.38 to -0.17], Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: CP-690,550 5 mg vs Placebo; LS Mean Difference and corresponding 95% CI was calculated using a mixed effect repeated measure model with treatment, visit, treatment by visit interaction, and geographic region as fixed effects and participants as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Step-down procedure: For the comparison of 5 mg to placebo to be statistically significant in this measure, the comparison of 10 mg to placebo as well as the comparison of 5 mg to placebo in ACR20 had to be statistically significant; LS Mean Difference = -0.25, 95% CI 2-sided [-0.36 to -0.15], Standard Error of Mean 0.05

3. Primary Outcome: Percentage of Participants With Disease Activity Score Based on 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) Less Than 2.6 at Month 3
Description: DAS28-4 (ESR) was calculated from SJC and TJC using 28 joints count, erythrocyte sedimentation rate (ESR)(millimeter/hour [mm/hour]) and patient's global assessment (PtGA) of disease activity (participant rated arthritis activity assessment). Total score range:0-9.4, higher score=more disease activity. DAS28-4 (ESR) less than or equal to (<=)3.2 implied low disease activity, greater than (>)3.2 to 5.1 implied moderate to high disease activity, less than (<)2.6=remission. For comparison of CP-690,550 with placebo, placebo sequences were combined into single reporting group for Month 3 analysis.
Time Frame: Month 3
Population: FAS included all randomized participants who received at least 1 dose of study treatment and had at least 1 post-baseline measurement. Missing values due to participant dropping due to any reason were imputed using NRI. Here 'N' (Number of Participants Analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 119 | 125 | 120
percentage of participants | 6.72 | 11.20 | 1.67
Statistical Analysis 1: Comparison: CP-690,550 10 mg vs Placebo; Normal approximation for the difference in binomial proportions was used to test the superiority of CP-690,550 10 mg to placebo and 2-sided 95% CI was evaluated for the difference in percentages; Test type: Superiority or Other; p = 0.0017, Normal Approximation — A step-down procedure was used to control for multiple comparisons. For the comparison of 10 mg to placebo to be statistically significant in this measure, the comparison of 10 mg to placebo in HAQ-DI had to be statistically significant; Percentage Difference = 9.53, 95% CI 2-sided [3.54 to 15.51], Standard Error of Mean 3.05
Statistical Analysis 2: Comparison: CP-690,550 5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0496, Normal Approximation — Step-down procedure: For the comparison of 5 mg to placebo to be statistically significant in this measure, the comparison of 10 mg to placebo as well as comparison of 5 mg to placebo in HAQ-DI had to be statistically significant; Percentage Difference = 5.05, 95% CI 2-sided [0.00 to 10.10], Standard Error of Mean 2.57

4. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Week 2 and Month 1
Description: ACR20 response: >=20% improvement in TJC; >=20% improvement in SJC; and >= 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Week 2, Month 1
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 132 | 133 | 131
percentage of participants
  Week 2 | 27.69 | 32.81 | 16.67
  Month 1 | 42.42 | 44.36 | 27.48

5. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Month 4.5 and 6
Description: ACR20 response: >=20% improvement in TJC; >=20% improvement in SJC; and >=20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Month 4.5, 6
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 132 | 133 | 66 | 65
percentage of participants
  Month 4.5 | 54.55 | 47.37 | 50.00 | 46.15
  Month 6 | 51.52 | 54.89 | 45.45 | 40.00

6. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response at Week 2, Month 1 and 3
Description: ACR50 response: >= 50% improvement in TJC or SJC and 50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Week 2, Month 1, 3
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 132 | 133 | 131
percentage of participants
  Week 2 | 7.69 | 5.47 | 1.59
  Month 1 | 12.88 | 17.29 | 6.11
  Month 3 | 26.52 | 27.82 | 8.40

7. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response at Month 4.5 and 6
Description: as for outcome 6
Time Frame: Month 4.5 and 6
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 132 | 133 | 66 | 65
percentage of participants
  Month 4.5 | 28.79 | 28.57 | 30.30 | 20.00
  Month 6 | 37.12 | 30.08 | 28.79 | 20.00

8. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response at Week 2, Month 1 and 3
Description: ACR70 response: >=70% improvement in TJC or SJC and 70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Week 2, Month 1, 3
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 132 | 133 | 131
percentage of participants
  Week 2 | 2.31 | 2.34 | 0.00
  Month 1 | 7.58 | 6.77 | 0.00
  Month 3 | 13.64 | 10.53 | 1.53

9. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response at Month 4.5 and 6
Description: as for outcome 8
Time Frame: Month 4.5, 6
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 132 | 133 | 66 | 65
percentage of participants
  Month 4.5 | 10.61 | 12.78 | 12.12 | 7.69
  Month 6 | 15.91 | 15.79 | 10.61 | 9.23

10. Secondary Outcome: Disease Activity Score Based on 28-Joints Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP]) at Baseline, Week 2, Month 1 and 3
Description: DAS28-3 (CRP) was calculated from the SJC and TJC using the 28 joints count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) <=3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity, and DAS28-3 (CRP) <2.6 = remission.
Time Frame: Baseline, Week 2, Month 1, 3
Population: FAS included all randomized participants who received at least 1 dose of study treatment and had at least 1 post-baseline measurement. Here 'n' signifies participants who were evaluable at specified time points for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 133 | 134 | 132
units on a scale
  Baseline (n=133,134,132) | 5.38 (1.00) | 5.31 (0.90) | 5.39 (0.95)
  Week 2 (n=127,125,124) | 4.46 (1.23) | 4.13 (1.04) | 5.10 (1.13)
  Month 1 (n=123,123,123) | 4.14 (1.27) | 3.92 (1.19) | 4.92 (1.20)
  Month 3 (n=118,124,118) | 3.74 (1.31) | 3.45 (1.32) | 4.78 (1.34)

11. Secondary Outcome: Disease Activity Score Based on 28-Joints Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP]) at Month 4.5 and 6
Description: DAS28-3 (CRP) was calculated from the SJC and TJC using the 28 joints count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) <= 3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity, and DAS28-3 (CRP) <2.6 = remission.
Time Frame: Month 4.5, 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 112 | 113 | 56 | 51
units on a scale
  Month 4.5 (n=112,113,56,51) | 3.43 (1.25) | 3.30 (1.37) | 3.57 (1.15) | 3.69 (1.15)
  Month 6 (n=100,102,51,48) | 3.36 (1.24) | 3.07 (1.18) | 3.46 (1.13) | 3.68 (1.19)

12. Secondary Outcome: Disease Activity Score Based on 28-Joints Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) at Baseline and Month 3
Description: DAS28-4 (ESR) was calculated from SJC and TJC using 28 joints count, ESR (mm/hour) and PtGA of disease activity (participant rated arthritis activity assessment). Total score range: 0-9.4, higher score=more disease activity. DAS28-4 (ESR) <= 3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity, and DAS28-4 (ESR) <2.6 = remission.
Time Frame: Baseline, Month 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 126 | 128 | 130
units on a scale
  Baseline (n=126,128,130) | 6.48 (1.03) | 6.40 (0.89) | 6.47 (0.98)
  Month 3 (n=112,121,110) | 4.58 (1.39) | 4.26 (1.48) | 5.56 (1.45)

13. Secondary Outcome: Disease Activity Score Based on 28-Joints Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) at Month 6
Description: as for outcome 12
Time Frame: Month 6
Population: FAS included all randomized participants who received at least 1 dose of study treatment and had at least 1 post-baseline measurement. Here 'N' (Number of Participants Analyzed) signifies participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 100 | 100 | 49 | 47
units on a scale | 3.99 (1.41) | 3.70 (1.25) | 4.07 (1.26) | 4.39 (1.27)

14. Secondary Outcome: Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 2, Month 1 and 3
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; common activities over past week. Each item scored on 4-point scale from 0-3:0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as sum of domain scores and divided by number of domains answered. Total possible score range 0-3:0=least difficulty and 3=extreme difficulty.
Time Frame: Week 2, Month 1, 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 130 | 128 | 125
units on a scale
  Week 2 (n=130,128,125) | 1.38 (0.71) | 1.28 (0.58) | 1.49 (0.63)
  Month 1 (n=123,123,123) | 1.37 (0.68) | 1.19 (0.65) | 1.38 (0.72)
  Month 3 (n=118,125,118) | 1.20 (0.72) | 1.10 (0.66) | 1.44 (0.72)

15. Secondary Outcome: Health Assessment Questionnaire-Disability Index (HAQ-DI) at Month 4.5 and 6
Description: as for outcome 14
Time Frame: Month 4.5, 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 112 | 114 | 57 | 53
units on a scale
  Month 4.5 (n=112,114,57,53) | 1.19 (0.69) | 1.10 (0.70) | 1.08 (0.60) | 1.26 (0.75)
  Month 6 (n=104,103,51,49) | 1.10 (0.70) | 1.02 (0.65) | 1.00 (0.59) | 1.29 (0.72)

16. Secondary Outcome: Patient Assessment of Arthritis Pain at Baseline, Week 2, Month 1 and 3
Description: Participants rated the severity of arthritis pain on a 0 to 100 millimeter (mm) Visual Analog Scale (VAS), where 0 mm = no pain and 100 mm = most severe pain.
Time Frame: Baseline, Week 2, Month 1, 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 130 | 128 | 131
units on a scale
  Baseline (n=127,128,131) | 65.73 (22.79) | 60.10 (23.16) | 60.74 (23.50)
  Week 2 (n=130,128,125) | 49.79 (26.60) | 42.35 (22.11) | 55.88 (23.85)
  Month 1 (n=124,122,123) | 45.59 (26.02) | 39.09 (24.05) | 52.29 (25.65)
  Month 3 (n=119,124,116) | 38.91 (27.11) | 37.72 (26.99) | 53.40 (26.52)

17. Secondary Outcome: Patient Assessment of Arthritis Pain at Month 4.5 and 6
Description: Participants rated the severity of arthritis pain on a 0 to 100 mm VAS, where 0 mm = no pain and 100 mm = most severe pain.
Time Frame: Month 4.5, 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 112 | 115 | 56 | 53
units on a scale
  Month 4.5 (n=112,115,56,53) | 38.93 (26.40) | 35.01 (24.60) | 33.11 (23.44) | 40.62 (26.67)
  Month 6 (n=104,103,51,49) | 34.38 (25.33) | 29.56 (22.77) | 31.37 (24.76) | 40.71 (25.88)

18. Secondary Outcome: Patient Global Assessment (PtGA) of Arthritis Pain at Baseline, Week 2, Month 1 and 3
Description: Participants answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using a 0 - 100 mm VAS, where 0 mm = very well and 100 mm = very poorly.
Time Frame: Baseline, Week 2, Month 1, 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 130 | 128 | 131
units on a scale
  Baseline (n=127,128,131) | 64.69 (23.22) | 58.79 (23.59) | 61.87 (22.92)
  Week 2 (n=130,128,124) | 48.24 (25.54) | 41.75 (21.79) | 57.70 (23.77)
  Month 1 (n=124,123,123) | 44.86 (25.62) | 38.35 (23.38) | 51.39 (26.01)
  Month 3 (n=119,125,118) | 41.23 (27.06) | 37.23 (25.65) | 52.85 (25.64)

19. Secondary Outcome: Patient Global Assessment (PtGA) of Arthritis Pain at Month 4.5 and 6
Description: as for outcome 18
Time Frame: Month 4.5, 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 112 | 115 | 56 | 53
units on a scale
  Month 4.5 (n=112,115,56,53) | 37.40 (24.65) | 36.01 (25.46) | 34.38 (23.47) | 38.79 (26.17)
  Month 6 (n=104,103,51,49) | 34.59 (24.82) | 31.25 (23.25) | 34.88 (23.84) | 38.61 (22.27)

20. Secondary Outcome: Physician Global Assessment of Arthritis at Baseline, Week 2, Month 1 and 3
Description: Physician Global Assessment of Arthritis was measured on a 0 to 100 mm VAS, where 0 mm = very good and 100 mm = very bad.
Time Frame: Baseline, Week 2, Month 1, 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 129 | 128 | 131
units on a scale
  Baseline (n=126,128,131) | 65.38 (18.21) | 58.68 (19.42) | 64.36 (16.70)
  Week 2 (n=129,128,123) | 46.51 (23.38) | 41.29 (20.58) | 51.36 (21.87)
  Month 1 (n=123,122,123) | 39.88 (22.19) | 36.28 (21.52) | 47.67 (20.84)
  Month 3 (n=117,124,116) | 34.94 (25.22) | 30.64 (22.20) | 44.08 (23.53)

21. Secondary Outcome: Physician Global Assessment of Arthritis at Month 4.5 and 6
Description: as for outcome 20
Time Frame: Month 4.5, 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 110 | 114 | 55 | 53
units on a scale
  Month 4.5 (n=110,114,55,53) | 27.50 (18.87) | 26.12 (22.28) | 28.67 (19.77) | 28.17 (21.50)
  Month 6 (n=101,101,51,48) | 24.17 (18.55) | 19.65 (17.15) | 23.55 (18.30) | 23.75 (16.20)

22. Secondary Outcome: 36-Item Short-Form Health Survey (SF-36) at Baseline, Week 2, Month 1 and 3
Description: SF-36 is a standardized survey evaluating 8 domains (of 2 components; physical and mental) of functional health and well being: physical and social functioning, physical and emotional role (role-physical, role-emotional) limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
Time Frame: Baseline, Week 2, Month 1, 3
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 133 | 134 | 132
units on a scale
  Baseline:Physical Functioning (n=133,134,132) | 30.54 (10.76) | 31.61 (8.58) | 28.32 (9.30)
  Baseline:Role Physical (n=133,134,132) | 33.66 (10.21) | 34.08 (9.67) | 32.53 (9.66)
  Baseline:Bodily Pain (n=133,134,132) | 31.09 (8.13) | 32.55 (7.45) | 31.95 (7.70)
  Baseline:General Health (n=133,134,132) | 35.84 (9.50) | 37.73 (9.18) | 34.82 (8.67)
  Baseline:Vitality (n=133,134,132) | 39.71 (9.87) | 40.11 (10.26) | 38.41 (10.77)
  Baseline:Social Functioning (n=133,134,132) | 37.40 (13.10) | 39.47 (12.11) | 35.95 (12.39)
  Baseline:Role Emotional (n=133,134,132) | 37.58 (14.08) | 36.75 (13.58) | 35.52 (14.22)
  Baseline:Mental Health (n=133,134,132) | 40.66 (11.63) | 41.91 (11.99) | 39.69 (12.66)
  Baseline:Physical Component Score(n=133,134,132) | 30.72 (9.29) | 32.13 (7.58) | 29.98 (7.99)
  Baseline: Mental Component Score (n=133,134,132) | 42.82 (12.69) | 43.24 (12.81) | 41.34 (13.25)
  Week 2:Physical Functioning (n=130,128,125) | 33.28 (11.06) | 34.25 (9.30) | 30.25 (10.30)
  Week 2:Role Physical (n=130,128,125) | 36.71 (10.23) | 38.45 (9.04) | 36.05 (10.48)
  Week 2:Bodily Pain (n=130,128,125) | 37.01 (9.34) | 38.42 (7.70) | 33.77 (7.80)
  Week 2:General Health (n=130,128,125) | 37.38 (8.52) | 38.57 (8.61) | 35.85 (8.76)
  Week 2:Vitality (n=130,128,125) | 43.02 (10.18) | 43.89 (10.71) | 41.11 (10.62)
  Week 2:Social Functioning (n=130,128,125) | 41.18 (12.79) | 42.29 (11.29) | 38.08 (12.18)
  Week 2:Role Emotional (n=130,128,125) | 40.54 (12.94) | 40.62 (11.99) | 37.69 (13.49)
  Week 2:Mental Health (n=130,128,125) | 43.72 (11.48) | 44.25 (11.19) | 42.07 (12.31)
  Week 2:Physical Component Score (n=130,128,125) | 34.04 (9.51) | 35.69 (7.74) | 31.99 (8.58)
  Week 2:Mental Component Score (n=130,128,125) | 45.77 (11.93) | 45.98 (11.95) | 43.57 (12.74)
  Month 1:Physical Functioning (n=124,123,123) | 33.56 (11.14) | 35.64 (10.06) | 31.01 (10.15)
  Month 1: Role Physical (n=124,123,123) | 38.25 (10.06) | 39.59 (9.98) | 36.33 (10.56)
  Month 1:Bodily Pain(n=124,123,123) | 37.50 (9.45) | 40.02 (8.42) | 35.35 (8.77)
  Month 1:General Health (n=124,123,123) | 38.09 (9.32) | 39.82 (9.25) | 36.64 (8.75)
  Month 1:Vitality (n=124,123,123) | 44.33 (9.35) | 45.65 (11.47) | 41.85 (11.50)
  Month 1:Social Functioning (n=124,123,123) | 40.96 (11.62) | 44.12 (11.65) | 39.00 (12.49)
  Month 1:Role Emotional (n=124,123,123) | 41.05 (13.23) | 40.84 (12.86) | 38.87 (12.84)
  Month 1:Mental Health (n=124,123,123) | 44.13 (11.68) | 46.18 (11.64) | 42.89 (11.92)
  Month 1:Physical Component Score (n=124,123,123) | 34.88 (9.24) | 37.07 (8.40) | 32.72 (9.18)
  Month 1:Mental Component Score (n=124,123,123) | 46.13 (11.94) | 47.28 (12.47) | 44.53 (12.42)
  Month 3:Physical Functioning (n=118,125,117) | 34.78 (11.43) | 36.70 (10.56) | 30.54 (10.67)
  Month 3: Role Physical (n=118,125,117) | 38.40 (10.49) | 40.19 (10.95) | 35.09 (10.66)
  Month 3:Bodily Pain (n=118,125,117) | 39.25 (9.78) | 40.93 (9.67) | 34.26 (9.62)
  Month 3:General Health (n=118,125,117) | 39.22 (9.78) | 40.21 (9.46) | 35.30 (9.30)
  Month 3:Vitality (n=118,125,117) | 45.23 (10.89) | 46.23 (11.73) | 40.30 (11.71)
  Month 3:Social Functioning (n=118,125,117) | 41.91 (12.37) | 44.49 (11.21) | 37.74 (12.12)
  Month 3:Role Emotional (n=118,125,116) | 41.21 (12.57) | 41.84 (12.67) | 36.16 (14.50)
  Month 3:Mental Health (n=118,125,117) | 44.58 (11.95) | 45.83 (11.59) | 40.89 (12.46)
  Month 3:Physical Component Score (n=118,125,116) | 36.18 (9.96) | 38.01 (9.35) | 32.38 (9.35)
  Month 3:Mental Component Score (n=118,125,116) | 46.40 (11.87) | 47.37 (12.01) | 41.91 (12.85)

23. Secondary Outcome: 36-Item Short-Form Health Survey (SF-36) at Month 6
Description: as for outcome 22
Time Frame: Month 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 104 | 103 | 51 | 49
units on a scale
  Month 6:Physical Functioning | 35.62 (11.63) | 38.47 (10.14) | 35.00 (10.31) | 33.97 (10.58)
  Month 6: Role Physical | 40.72 (9.95) | 43.51 (11.21) | 39.54 (10.55) | 38.02 (9.81)
  Month 6:Bodily Pain | 41.53 (9.61) | 43.63 (9.27) | 42.40 (10.22) | 39.60 (9.01)
  Month 6:General Health | 39.49 (9.54) | 41.68 (10.35) | 38.95 (9.51) | 37.89 (8.45)
  Month 6:Vitality | 46.49 (9.82) | 47.59 (10.93) | 45.09 (12.26) | 44.26 (8.73)
  Month 6:Social Functioning | 44.05 (10.93) | 44.66 (11.92) | 43.33 (12.27) | 40.38 (11.11)
  Month 6:Role Emotional | 42.36 (13.34) | 45.06 (12.27) | 41.07 (13.18) | 39.53 (12.93)
  Month 6:Mental Health | 45.29 (12.12) | 47.48 (11.61) | 44.85 (14.61) | 46.19 (9.65)
  Month 6:Physical Component Score | 37.78 (9.20) | 40.21 (9.24) | 37.84 (9.59) | 35.43 (8.69)
  Month 6:Mental Component Score | 47.41 (12.32) | 48.83 (12.65) | 46.17 (15.06) | 46.03 (11.52)

24. Secondary Outcome: Medical Outcomes Study Sleep Scale (MOS-SS) at Baseline, Week 2, Month 1 and 3
Description: Participant-rated 12-item questionnaire to assess constructs of sleep over past week; 7 subscales:sleep disturbance,snoring,awakened short of breath,sleep adequacy,somnolence (range:0-100);sleep quantity (range:0-24),optimal sleep(yes/no), and 9 item index measures of sleep disturbance provide composite scores:sleep problem summary,overall sleep problem.Except adequacy,optimal sleep and quantity,higher scores=more impairment.Scores transformed(actual raw score[RS] minus lowest possible score divided by possible RS range*100);total score range:0-100;higher score=more intensity of attribute.
Time Frame: Baseline, Week 2, Month 1, 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 133 | 133 | 130
units on a scale
  Baseline: Sleep Problem Summary (n=133,132,129) | 40.55 (21.13) | 39.87 (18.03) | 44.65 (20.56)
  Baseline: Overall Sleep Problem (n=133,132,129) | 43.10 (21.00) | 41.57 (17.88) | 46.08 (20.73)
  Baseline: Sleep Adequacy (n=133,133,129) | 46.39 (27.89) | 43.16 (25.89) | 39.53 (27.95)
  Baseline: Awakened Short of Breath (n=133,133,130) | 16.99 (24.56) | 19.10 (24.10) | 21.54 (26.19)
  Baseline: Sleep Disturbance (n=133,133,129) | 47.43 (28.39) | 43.20 (24.83) | 47.98 (27.00)
  Baseline: Sleep Quantity (n=132,131,129) | 6.47 (1.55) | 6.44 (1.35) | 6.33 (1.46)
  Baseline: Snoring (n=131,131,127) | 42.14 (31.89) | 37.10 (33.75) | 40.00 (33.62)
  Baseline: Somnolence (n=133,132,129) | 36.39 (22.47) | 34.19 (22.83) | 38.55 (23.60)
  Week 2: Sleep Problem Summary (n=129,127,125) | 36.87 (20.84) | 37.03 (18.97) | 40.35 (20.10)
  Week 2: Overall Sleep Problem (n=129,127,124) | 38.04 (20.78) | 37.69 (18.83) | 41.47 (20.01)
  Week 2: Sleep Adequacy (n=129,127,125) | 48.06 (28.70) | 44.17 (28.35) | 42.72 (26.77)
  Week 2: Awakened Short of Breath (n=129,127,125) | 17.83 (25.28) | 17.32 (21.58) | 18.72 (25.75)
  Week 2: Sleep Disturbance (n=129,127,125) | 39.59 (28.24) | 36.41 (22.89) | 42.28 (26.45)
  Week 2: Sleep Quantity (n=129,127,124) | 6.40 (1.57) | 6.68 (1.41) | 6.48 (1.75)
  Week 2: Snoring (n=128,125,122) | 36.25 (34.21) | 35.84 (34.48) | 40.49 (32.67)
  Week 2: Somnolence (n=129,127,124) | 31.78 (21.85) | 32.18 (23.47) | 36.45 (23.18)
  Month 1: Sleep Problem Summary (n=124,123,123) | 36.21 (20.69) | 34.53 (20.08) | 37.37 (20.42)
  Month 1: Overall Sleep Problem (n=124,123,123) | 37.23 (20.70) | 35.40 (19.94) | 38.79 (20.58)
  Month 1: Sleep Adequacy (n=124,123,123) | 49.84 (28.31) | 48.13 (29.35) | 49.11 (28.86)
  Month 1: Awakened Short of Breath (n=124,123,123) | 15.81 (21.53) | 15.45 (23.16) | 19.84 (26.30)
  Month 1: Sleep Disturbance (n=124,123,123) | 39.12 (28.16) | 34.82 (25.12) | 39.64 (26.26)
  Month 1: Sleep Quantity (n=124,123,123) | 6.59 (1.34) | 6.80 (1.43) | 6.43 (1.42)
  Month 1: Snoring (n=124,122,120) | 36.13 (33.42) | 34.10 (32.80) | 41.50 (33.12)
  Month 1: Somnolence (n=124,123,123) | 30.91 (22.30) | 30.84 (23.97) | 34.91 (23.67)
  Month 3: Sleep Problem Summary (n=117,125,117) | 36.81 (21.10) | 35.68 (19.36) | 40.14 (20.20)
  Month 3: Overall Sleep Problem (n=117,125,117) | 37.23 (20.72) | 36.08 (19.40) | 42.00 (20.41)
  Month 3: Sleep Adequacy (n=118,125,117) | 48.64 (30.32) | 48.56 (29.04) | 43.68 (27.47)
  Month 3: Awakened Short of Breath (n=118,125,117) | 18.14 (23.68) | 19.68 (24.09) | 17.95 (24.27)
  Month 3: Sleep Disturbance (n=118,125,117) | 38.44 (28.37) | 34.61 (23.21) | 43.27 (26.45)
  Month 3: Sleep Quantity (n=117,124,117) | 6.58 (1.50) | 6.71 (1.42) | 6.27 (1.49)
  Month 3: Snoring (n=118,123,117) | 36.44 (32.83) | 36.26 (32.63) | 41.37 (31.92)
  Month 3: Somnolence (n=117,125,117) | 30.14 (23.53) | 31.31 (23.68) | 36.47 (23.10)

25. Secondary Outcome: Medical Outcomes Study Sleep Scale (MOS-SS) at Month 6
Description: as for outcome 24
Time Frame: Month 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 104 | 102 | 49 | 49
units on a scale
  Month 6: Sleep Problem Summary | 35.32 (21.46) | 32.03 (18.42) | 38.78 (20.81) | 35.35 (19.05)
  Month 6: Overall Sleep Problem | 35.75 (20.68) | 32.92 (18.33) | 39.73 (20.85) | 36.02 (18.45)
  Month 6: Sleep Adequacy | 50.48 (30.64) | 52.75 (28.46) | 43.47 (30.99) | 50.42 (26.89)
  Month 6: Awakened Short of Breath | 16.73 (24.15) | 14.12 (22.62) | 18.37 (21.54) | 17.92 (21.13)
  Month 6: Sleep Disturbance | 36.84 (26.19) | 33.88 (23.51) | 40.92 (26.89) | 35.10 (25.26)
  Month 6: Sleep Quantity | 6.56 (1.45) | 6.93 (1.29) | 6.27 (1.29) | 6.80 (1.26)
  Month 6: Snoring | 34.62 (31.80) | 35.84 (31.79) | 37.96 (31.95) | 38.75 (32.59)
  Month 6: Somnolence | 29.74 (22.24) | 26.14 (19.40) | 30.61 (22.56) | 33.19 (20.09)

26. Secondary Outcome: Number of Participants With Optimal Sleep Assessed Using Medical Outcomes Study Sleep Scale (MOS-SS) at Baseline, Week 2, Month 1, and 3
Description: MOS-SS: participant-rated 12 item questionnaire to assess constructs of sleep over past week. It included 7 subscales: sleep disturbance, snoring, awakened short of breath, sleep adequacy, somnolence, sleep quantity and optimal sleep. Participants responded whether their sleep was optimal or not optimal by choosing yes or no. Number of participants with optimal sleep is reported.
Time Frame: Baseline, Week 2, Month 1, 3
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 133 | 134 | 132
participants
  Baseline (n= 133, 134, 132) | 53 | 59 | 48
  Week 2 (n= 130, 128, 126) | 52 | 62 | 50
  Month 1 (n= 124, 123, 124) | 59 | 58 | 53
  Month 3 (n= 118, 125, 118) | 53 | 56 | 47

27. Secondary Outcome: Number of Participants With Optimal Sleep Assessed Using Medical Outcomes Study Sleep Scale (MOS-SS) at Month 6
Description: as for outcome 26
Time Frame: Month 6
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 104 | 103 | 51 | 49
participants | 50 | 57 | 21 | 24

28. Secondary Outcome: Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale at Baseline and Month 3
Description: FACIT-Fatigue Scale (FS):13-item questionnaire, participant scored each item on a 5-point scale: 0 (not at all) to 4 (very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as 4 minus the participant's response. The sum of all responses resulted in the FACIT-FS for a total possible score of 0 (worse score) to 52 (better score). A higher score reflected an improvement in the participant's health status.
Time Frame: Baseline, Month 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 132 | 134 | 129
units on a scale
  Baseline (n=132,134,129) | 27.84 (11.12) | 29.48 (11.39) | 26.98 (11.52)
  Month 3 (n=118,125,117) | 33.30 (11.72) | 33.66 (12.27) | 27.93 (12.36)

29. Secondary Outcome: Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale at Month 6
Description: FACIT-FS:13-item questionnaire, participant scored each item on a 5-point scale: 0 (not at all) to 4 (very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as 4 minus the participant's response. The sum of all responses resulted in the FACIT-FS for a total possible score of 0 (worse score) to 52 (better score). A higher score reflected an improvement in the participant's health status.
Time Frame: Month 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 104 | 102 | 51 | 49
units on a scale | 34.69 (10.81) | 35.98 (11.55) | 33.57 (12.21) | 31.63 (10.16)

30. Secondary Outcome: Euro Quality of Life - 5 Dimensions (EQ-5D)- Health State Profile Utility Score at Baseline, Month 1 and 3
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state (confined to bed). Scoring formula developed by EuroQoL Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline, Month 1, 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 131 | 134 | 129
units on a scale
  Baseline (n=131,134,129) | 0.38 (0.34) | 0.47 (0.32) | 0.38 (0.33)
  Month 1 (n=122,121,120) | 0.56 (0.28) | 0.63 (0.24) | 0.49 (0.30)
  Month 3 (n=117,123,117) | 0.55 (0.30) | 0.62 (0.25) | 0.43 (0.35)

31. Secondary Outcome: Euro Quality of Life - 5 Dimensions (EQ-5D) - Health State Profile Utility Score at Month 6
Description: as for outcome 30
Time Frame: Month 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 104 | 101 | 51 | 49
units on a scale | 0.62 (0.28) | 0.68 (0.24) | 0.60 (0.24) | 0.55 (0.29)

32. Secondary Outcome: Work Productivity and Healthcare Resource Utilization (HCRU) at Baseline, Month 3
Description: Rheumatoid Arthritis (RA)-HCRU assessed healthcare usage during last 3 months for direct, indirect medical cost domains. Direct cost:visit to doctor,non-medical practitioner,nursing home,hospital,surgery,emergency room(ER) treatment,diagnostic tests, over-night stay,home healthcare services, aids/devices used. Indirect costs associated with functional disability:employment status,willingness to work,work disability due to RA,sick leave,part time work,ability to perform chores,chores done by family/friends/housekeeper. Assessment was based on 0 to 2-point scale;higher score=higher medical cost.
Time Frame: Baseline, Month 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 133 | 134 | 130
units on a scale
  Baseline: Seen any doctor (n=133,133,130) | 1.11 (0.31) | 1.09 (0.29) | 1.15 (0.35)
  Baseline: Treated in ER (n=133,134,130) | 1.89 (0.32) | 1.96 (0.19) | 1.93 (0.25)
  Baseline: Admitted for overnight stay (n=16,6,9) | 0.19 (0.54) | 0.17 (0.41) | 0.33 (0.71)
  Baseline: Hospitalization (n=133,134,130) | 1.97 (0.17) | 1.97 (0.17) | 1.95 (0.23)
  Baseline: Had outpatient surgeries (n=133,134,130) | 1.95 (0.21) | 1.97 (0.17) | 1.93 (0.25)
  Baseline:Non-study diagnostic tests(n=133,134,130) | 1.74 (0.44) | 1.75 (0.43) | 1.74 (0.44)
  Baseline: In nursing home (n=133,134,130) | 1.99 (0.09) | 1.99 (0.09) | 1.99 (0.09)
  Baseline: Home HC services (n=133,134,130) | 1.98 (0.12) | 1.99 (0.09) | 1.96 (0.19)
  Baseline: Home healthcare services (n=2,2,5) | 1.50 (0.71) | 0.50 (0.71) | 0.80 (0.84)
  Baseline:Required aids/devices (n=133,134,130) | 1.77 (0.42) | 1.86 (0.35) | 1.82 (0.39)
  Baseline: Seen NM practitioner (n=133,134,130) | 1.97 (0.17) | 1.96 (0.21) | 1.96 (0.19)
  Baseline: Currently employed (n=132,134,130) | 1.70 (0.46) | 1.66 (0.48) | 1.68 (0.47)
  Baseline: Feel well enough to work (n=84,78,83) | 1.85 (0.36) | 1.82 (0.39) | 1.82 (0.39)
  Baseline: Retired (n=85,80,86) | 1.49 (0.50) | 1.43 (0.50) | 1.49 (0.50)
  Baseline: Lost job/retired early (n=83,77,80) | 1.58 (0.50) | 1.69 (0.47) | 1.55 (0.50)
  Baseline: Unable to work due to RA (n=84,77,83) | 1.36 (0.48) | 1.48 (0.50) | 1.40 (0.49)
  Baseline: Work disabled due to RA (n=83,77,79) | 1.46 (0.50) | 1.55 (0.50) | 1.48 (0.50)
  Baseline: Sick leave due to RA (n=104,109,100) | 1.83 (0.38) | 1.80 (0.40) | 1.71 (0.46)
  Baseline: Performed part time work (n=103,108,100) | 1.94 (0.24) | 1.94 (0.25) | 1.88 (0.33)
  Baseline: Performed paid work (n=102,109,98) | 1.65 (0.48) | 1.63 (0.48) | 1.65 (0.48)
  Baseline: Unable to do chores (n=130,130,126) | 1.37 (0.48) | 1.42 (0.49) | 1.27 (0.45)
  Baseline: Chores by housekeeper (n=130,134,130) | 1.85 (0.36) | 1.86 (0.35) | 1.82 (0.39)
  Baseline: Chores by family/friends (n=131,134,130) | 1.44 (0.50) | 1.49 (0.50) | 1.48 (0.50)
  Month 3: Seen any doctor (n=117,125,117) | 1.23 (0.42) | 1.21 (0.41) | 1.21 (0.41)
  Month 3: Treated in ER (n=116,125,117) | 1.94 (0.24) | 1.94 (0.25) | 1.93 (0.25)
  Month 3: Admitted for overnight stay (n=7,8,8) | 0.29 (0.76) | 0.00 (0.00) | 0.13 (0.35)
  Month 3: Hospitalization (n=116,124,117) | 1.99 (0.09) | 2.00 (0.00) | 1.98 (0.13)
  Month 3: Had outpatient surgeries (n=116,125,117) | 1.94 (0.24) | 1.98 (0.15) | 1.97 (0.18)
  Month 3:Non study diagnostic tests (n=116,125,117) | 1.80 (0.40) | 1.82 (0.38) | 1.77 (0.42)
  Month 3: In nursing home (n=116,125,117) | 1.99 (0.09) | 1.99 (0.09) | 1.99 (0.09)
  Month 3: Home HC services (n=116,123,117) | 1.97 (0.16) | 1.99 (0.09) | 1.97 (0.16)
  Month 3: Required aids/devices (n=116,125,117) | 1.81 (0.39) | 1.91 (0.28) | 1.76 (0.43)
  Month 3: Seen NM practitioner (n=116,125,117) | 1.97 (0.18) | 1.97 (0.18) | 1.97 (0.18)
  Month 3: Currently employed (n=115,125,117) | 1.70 (0.46) | 1.62 (0.49) | 1.68 (0.47)
  Month 3: Feel well enough to work (n=68,67,70) | 1.82 (0.38) | 1.78 (0.42) | 1.83 (0.38)
  Month 3: Retired (n=68,66,72) | 1.56 (0.50) | 1.36 (0.48) | 1.53 (0.50)
  Month 3: Lost job/retired early (n=67,68,69) | 1.70 (0.46) | 1.69 (0.47) | 1.59 (0.49)
  Month 3: Unable to work due to RA (n=68,66,71) | 1.41 (0.50) | 1.53 (0.50) | 1.44 (0.50)
  Month 3: Work disabled due to RA (n=67,67,69) | 1.48 (0.50) | 1.57 (0.50) | 1.54 (0.50)
  Month 3: Sick leave due to RA (n=95,100,97) | 1.88 (0.32) | 1.86 (0.35) | 1.82 (0.38)
  Month 3: Performed part time work (n=96,100,96) | 1.96 (0.20) | 1.94 (0.24) | 1.94 (0.24)
  Month 3: Performed paid work (n=96,99,97) | 1.78 (0.42) | 1.69 (0.47) | 1.67 (0.47)
  Month 3: Unable to do chores (n=112,120,113) | 1.57 (0.50) | 1.63 (0.49) | 1.45 (0.50)
  Month 3: Chores by housekeeper (n=116,122,117) | 1.86 (0.35) | 1.89 (0.32) | 1.85 (0.35)
  Month 3: Chores by family/friends (n=116,122,116) | 1.55 (0.50) | 1.66 (0.48) | 1.53 (0.50)

33. Secondary Outcome: Work Productivity and Healthcare Resource Utilization (HCRU) at Month 6
Description: RA-HCRU assessed healthcare usage during last 3 months for direct, indirect medical cost domains. Direct cost: visit to doctor, non-medical practitioner, nursing home, hospital, surgery, emergency room(ER) treatment, diagnostic tests, over-night stay, home healthcare services, aids/devices used. Indirect costs associated with functional disability: employment status, willingness to work, work disability due to RA, sick leave, part time work, ability to perform chores, chores done by family/friends/housekeeper. Assessment was based on 0 to 2-point scale; higher score=higher medical cost.
Time Frame: Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 103 | 102 | 50 | 49
units on a scale
  Month 6: Seen any doctor (n=102,101,50,49) | 1.29 (0.46) | 1.22 (0.41) | 1.20 (0.40) | 1.27 (0.45)
  Month 6: Treated in ER (n=103,102,50,49) | 1.96 (0.19) | 1.93 (0.25) | 1.94 (0.24) | 1.98 (0.14)
  Month 6: Admitted for overnight stay (n=5,7,3,1) | 0.20 (0.45) | 0.00 (0.00) | 1.33 (1.15) | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Month 6: Hospitalization (n=102,102,50,49) | 1.98 (0.14) | 1.99 (0.10) | 1.96 (0.20) | 1.98 (0.14)
  Month 6:Had outpatient surgeries (n=103,102,50,49) | 2.00 (0.00) | 1.95 (0.22) | 1.96 (0.20) | 1.96 (0.20)
  Month 6:Non-study diagnostic test(n=103,102,50,49) | 1.85 (0.35) | 1.84 (0.37) | 1.74 (0.44) | 1.86 (0.35)
  Month 6: In nursing home (n=103,102,50,49) | 1.98 (0.14) | 2.00 (0.00) | 2.00 (0.00) | 1.96 (0.20)
  Month 6: Home HC services (n=101,102,50,49) | 2.00 (0.00) | 1.98 (0.14) | 2.00 (0.00) | 2.00 (0.00)
  Month 6: Required aids/devices (n=103,102,50,48) | 1.82 (0.39) | 1.91 (0.29) | 1.90 (0.30) | 1.83 (0.38)
  Month 6: Seen NM practitioner (n=103,102,50,49) | 1.99 (0.10) | 1.96 (0.20) | 1.98 (0.14) | 1.96 (0.20)
  Month 6: Currently employed (n=103,102,50,49) | 1.67 (0.47) | 1.63 (0.49) | 1.60 (0.49) | 1.71 (0.46)
  Month 6: Feel well enough to work (n=62,57,27,32) | 1.81 (0.40) | 1.68 (0.47) | 1.70 (0.47) | 1.88 (0.34)
  Month 6: Retired (n=62,56,28,31) | 1.45 (0.50) | 1.36 (0.48) | 1.43 (0.50) | 1.39 (0.50)
  Month 6: Lost job/retired early (n=62,54,27,32) | 1.71 (0.46) | 1.74 (0.44) | 1.59 (0.50) | 1.44 (0.50)
  Month 6: Unable to work due to RA (n=62,55,27,32) | 1.48 (0.50) | 1.67 (0.47) | 1.56 (0.51) | 1.41 (0.50)
  Month 6: Work disabled due to RA (n=61,53,27,32) | 1.57 (0.50) | 1.70 (0.46) | 1.56 (0.51) | 1.50 (0.51)
  Month 6: Sick leave due to RA (n=85,84,41,37) | 1.92 (0.28) | 1.88 (0.33) | 1.88 (0.33) | 1.86 (0.35)
  Month 6: Performed part time work (n=85,84,40,36) | 1.96 (0.19) | 1.95 (0.21) | 2.00 (0.00) | 1.92 (0.28)
  Month 6: Performed paid work (n=83,84,40,36) | 1.71 (0.46) | 1.75 (0.44) | 1.65 (0.48) | 1.64 (0.49)
  Month 6: Unable to do chores (n=101,98,49,48) | 1.65 (0.48) | 1.73 (0.44) | 1.51 (0.51) | 1.44 (0.50)
  Month 6: Chores by housekeeper (n=103,99,50,49) | 1.92 (0.27) | 1.91 (0.29) | 1.82 (0.39) | 1.90 (0.31)
  Month 6: Chores by family/friends (n=103,99,50,49) | 1.69 (0.47) | 1.77 (0.42) | 1.62 (0.49) | 1.55 (0.50)

34. Secondary Outcome: Number of Events Including Visits, Surgeries, Tests or Devices as Assessed Using RA-HCRU at Baseline and Month 3
Description: RA-HCRU assessed healthcare usage during previous 3 months for direct or indirect medical cost domains. Any RA/non-RA related number of events including visits to doctor, non-medical practitioner, hospital ER treatment, hospitalizations, number of surgeries, diagnostic tests, and devices/aids used were reported.
Time Frame: Baseline, Month 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of events
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 119 | 121 | 111
number of events
  Baseline: Doctor visit (n=119,121,111) | 5.07 (5.00) | 5.09 (5.10) | 4.58 (3.82)
  Baseline: NM practitioner visits (n=4,6,5) | 5.75 (4.35) | 4.83 (3.25) | 21.40 (29.75)
  Baseline: Hospital ER visit (n=14,5,9) | 1.79 (1.53) | 2.00 (1.73) | 1.22 (0.44)
  Baseline: Hospitalization (n=4,4,7) | 1.25 (0.50) | 1.00 (0.00) | 1.14 (0.38)
  Baseline: Outpatient surgery (n=6,4,8) | 1.17 (0.41) | 1.00 (0.00) | 1.00 (0.00)
  Baseline: Non-study diagnostic tests (n=34,32,32) | 1.85 (1.02) | 2.06 (1.72) | 1.69 (0.97)
  Baseline: RA related doctor visit (n=117,120,111) | 1.46 (0.91) | 1.18 (0.84) | 1.44 (0.93)
  Baseline: RA related ER visit (n=15,6,9) | 0.67 (0.90) | 0.67 (0.82) | 0.89 (0.93)
  Baseline: RA related diagnostic test (n=35,33,34) | 0.71 (0.83) | 0.79 (1.14) | 0.82 (0.76)
  Baseline: RA related hospitalization (n=4,5,7) | 0.75 (0.96) | 0.80 (1.10) | 0.86 (0.69)
  Baseline: RA related outpatient surgery (n=6,5,9) | 0.33 (0.82) | 0.80 (0.84) | 0.89 (0.93)
  Baselin:RA related NM visit (n=4,7,5) | 1.25 (0.96) | 0.57 (0.53) | 1.00 (1.00)
  Month 3: Doctor visit (n=89,99,93) | 3.30 (2.91) | 3.69 (3.73) | 4.04 (4.59)
  Month 3: NM practitioners visits (n=4,4,4) | 36.25 (40.25) | 5.00 (2.00) | 8.75 (10.63)
  Month 3: Hospital ER visit (n=7,8,8) | 1.00 (0.00) | 1.38 (1.06) | 1.38 (0.74)
  Month 3: Hospitalization (n=1,0,2) | 1.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 1.00 (0.00)
  Month 3: Outpatient surgery (n=7,3,4) | 1.14 (0.38) | 1.00 (0.00) | 1.00 (0.00)
  Month 3: Non-study diagnostic tests (n=22,22,26) | 1.82 (1.65) | 1.14 (0.35) | 1.62 (1.27)
  Month 3: RA related doctor visit (n=90,98,93) | 1.16 (1.08) | 0.82 (0.65) | 1.13 (0.92)
  Month 3: RA related ER visit (n=7,8,8) | 0.43 (0.79) | 0.00 (0.00) | 0.75 (1.39)
  Month 3: RA related diagnostic test (n=23,22,26) | 0.30 (0.47) | 0.23 (0.43) | 0.35 (0.56)
  Month 3: RA related hospitalization (n=1,0,2) | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 0.00 (0.00)
  Month 3:RA related outpatient surgery (n=7,3,4) | 0.43 (0.79) | 0.67 (1.15) | 1.00 (1.15)
  Month 3:RA related NM visit (n=4,4,4) | 0.75 (0.96) | 1.25 (0.96) | 1.25 (0.96)

35. Secondary Outcome: Number of Events Including Visits, Surgeries, Tests or Devices as Assessed Using RA-HCRU at Month 6
Description: as for outcome 34
Time Frame: Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of events
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 73 | 80 | 40 | 36
number of events
  Month 6: Doctor visit (n=73,80,39,36) | 3.26 (2.83) | 3.84 (4.25) | 3.64 (4.03) | 4.97 (6.73)
  Month 6: NM practitioner visit (n=1,4,1,2) | 5.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 15.50 (10.63) | 20.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 4.00 (0.00)
  Month 6: Hospital ER visit (n=4,7,3,1) | 1.25 (0.50) | 1.43 (0.79) | 1.67 (1.15) | 1.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Month 6: Hospitalization (n=2,1,2,1) | 2.00 (0.00) | 1.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 1.00 (0.00) | 1.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Month 6: Outpatient surgery (n=0,5,2,2) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 1.00 (0.00) | 2.50 (0.71) | 1.50 (0.71)
  Month 6: Non-study diagnostic test (n=15,16,13,7) | 2.07 (2.02) | 1.19 (0.54) | 1.85 (0.99) | 1.14 (0.38)
  Month 6: RA related doctor visit (n=73,80,40,36) | 1.10 (0.87) | 0.86 (0.76) | 0.85 (0.83) | 1.00 (0.96)
  Month 6: RA related ER visit (n=4,7,3,1) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Month 6: RA related diagnostic test (n=16,16,13,7) | 0.44 (0.73) | 0.00 (0.00) | 0.31 (0.85) | 0.29 (0.49)
  Month 6: RA related hospitalization (n=2,1,2,1) | 0.00 (0.00) | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 0.00 (0.00) | 2.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Month 6:RA related outpatient surgery (n=5,2,0,2) | 0.00 (0.00) | 2.00 (0.00) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 0.00 (0.00)
  Month6:RA related NM practitioner visit(n=1,4,1,2) | 1.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 2.00 (1.63) | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 1.00 (1.41)

36. Secondary Outcome: Number of Days as Assessed Using RA-HCRU at Baseline and Month 3
Description: RA-HCRU assessed healthcare usage during previous 3 months for direct or indirect medical cost domains. Any RA or non-RA related number of days spent in hospital, nursing home, aids/devices used, on sick leave, work per week, performed part time work, performed paid work, chores done by housekeeper and chores done by family/friends were reported.
Time Frame: Baseline, Month 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 71 | 65 | 66
days
  Baseline: Hospital length of stay (n=4,4,7) | 1.75 (0.96) | 7.00 (7.57) | 5.43 (3.78)
  Baseline: Days in nursing home (n=1,1,1) | 2.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 28.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 28.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Baseline: Days devices/aids used (n=31,18,24) | 122.94 (139.56) | 100.28 (122.82) | 94.63 (86.62)
  Baseline: Days of work per week (n=39,46,41) | 4.67 (1.24) | 4.83 (1.29) | 4.90 (1.18)
  Baseline: Chores by housekeeper (n=20,18,24) | 13.35 (20.32) | 20.56 (32.53) | 15.88 (23.45)
  Baseline: Chores by family/friend (n=71,65,66) | 27.55 (31.88) | 26.31 (32.27) | 27.38 (30.75)
  Baseline: Days on sick leave (n=17,22,28) | 19.76 (25.59) | 13.09 (16.15) | 23.71 (31.28)
  Baseline: Days of part time work (n=6,6,11) | 41.33 (40.41) | 6.83 (4.96) | 12.36 (16.20)
  Baseline: Paid work, bothered by RA (n=36,40,32) | 50.72 (63.36) | 39.75 (32.85) | 31.00 (30.79)
  Baseline: RA related devices/aids used (31,20,24) | 2.06 (1.59) | 1.75 (1.48) | 1.79 (0.88)
  Month 3: Hospital length of stay (n=1,0,2) | 12.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 11.00 (12.73)
  Month 3: Days in nursing home (n=1,1,1) | 9.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 21.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 21.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Month 3: Days devices/aids used (n=21,10,26) | 113.24 (102.65) | 264.10 (429.48) | 73.85 (70.60)
  Month 3: Days of work per week (n=33,47,37) | 4.94 (1.09) | 4.89 (1.09) | 4.65 (1.06)
  Month 3: Chores by housekeeper (n=15,14,17) | 13.00 (16.76) | 16.93 (31.22) | 10.12 (12.84)
  Month 3: Chores by family/friend (n=50,41,52) | 27.30 (31.13) | 24.24 (32.54) | 25.19 (36.03)
  Month 3: Days on sick leave (n=11,13,16) | 22.09 (28.51) | 6.62 (4.94) | 13.69 (20.16)
  Month 3: Days of part time work (n=4,4,5) | 8.25 (9.46) | 9.25 (7.89) | 8.20 (11.12)
  Month 3: Paid work, bothered by RA (n=19,29,28) | 26.58 (30.30) | 17.76 (23.98) | 30.54 (30.39)
  Month 3: RA related devices/aids used (22,11,27) | 2.09 (1.31) | 3.00 (4.45) | 2.04 (1.26)

37. Secondary Outcome: Number of Days as Assessed Using RA-HCRU at Month 6
Description: as for outcome 36
Time Frame: Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 83 | 84 | 40 | 36
days
  Month 6: Hospital length of stay (n=2,1,2,1) | 32.00 (33.94) | 3.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 25.00 (21.21) | 24.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Month 6: Days in nursing home (n=2,0,0,2) | 21.50 (0.71) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 13.50 (2.12)
  Month 6: Days devices/aids used (n=18,7,5,8) | 141.28 (105.31) | 68.43 (30.12) | 182.40 (87.11) | 75.00 (79.33)
  Month 6: Days of work per week (n=34,36,20,14) | 4.62 (1.33) | 4.97 (1.00) | 4.85 (0.99) | 4.71 (1.49)
  Month 6: Chores by housekeeper (n=8,9,9,5) | 12.75 (13.21) | 24.89 (36.09) | 9.22 (10.73) | 7.80 (4.55)
  Month 6: Chores by family/friend (n=32,23,18,19) | 28.91 (32.10) | 18.83 (26.97) | 19.33 (24.14) | 17.63 (26.46)
  Month 6: Days on sick leave (n=7,10,5,5) | 21.00 (31.86) | 10.40 (14.49) | 9.20 (11.17) | 42.60 (44.81)
  Month 6: Days of part time work (n=3,3,0,3) | 5.67 (8.08) | 9.33 (5.03) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 21.33 (33.49)
  Month 6: Paid work, bothered by RA (n=21,19,12,11) | 25.00 (32.76) | 14.95 (20.85) | 22.17 (31.98) | 19.64 (21.73)
  Month 6: RA related devices/aids used (19,8,5,8) | 2.05 (1.22) | 1.13 (0.64) | 2.20 (0.84) | 1.63 (1.19)

38. Secondary Outcome: Number of Hours Per Day as Assessed RA-HCRU at Baseline and Month 3
Description: RA-HCRU assessed healthcare usage during previous 3 months for direct or indirect medical cost domains. Any RA or non-RA related number of hours spent per day for home healthcare services, chores done by housekeeper, chores done by family or friends, hours affected per day and average number of hours missed work per day were reported.
Time Frame: Baseline, Month 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 71 | 63 | 66
hours per day
  Baseline: Home healthcare services (n=2,1,4) | 5.00 (4.24) | 3.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 7.25 (11.18)
  Baseline: Work done (n=39,45,41) | 9.41 (8.52) | 8.18 (7.18) | 8.98 (7.35)
  Baseline: Chores by housekeeper (n=19,18,23) | 4.68 (3.23) | 3.83 (1.54) | 4.78 (2.37)
  Baseline: Chores by family/friend (n=71,63,66) | 2.85 (1.89) | 4.44 (11.21) | 3.42 (2.61)
  Baseline: Missed work due to RA (n=6,6,11) | 2.67 (1.97) | 3.17 (2.23) | 7.55 (7.31)
  Baseline: RA related home HC services (n=2,2,5) | 1.50 (0.71) | 0.50 (0.71) | 0.80 (0.84)
  Month 3: Home healthcare services (n=3,1,3) | 4.00 (3.46) | 2.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 9.33 (12.70)
  Month 3: Work done (n=34,46,37) | 7.97 (4.72) | 9.20 (8.52) | 7.76 (1.98)
  Month 3: Chores by housekeeper (n=15,14,17) | 4.00 (2.20) | 3.71 (1.14) | 5.41 (5.26)
  Month 3: Chores by family/friend (n=50,41,49) | 3.50 (3.72) | 2.83 (2.57) | 4.00 (5.34)
  Month 3: Missed work due to RA (n=4,4,5) | 3.00 (2.00) | 6.25 (6.18) | 7.80 (9.12)
  Month 3: RA related home HC services (n=3,1,3) | 1.33 (0.58) | 1.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 1.67 (0.58)

39. Secondary Outcome: Number of Hours Per Day as Assessed RA-HCRU at Month 6
Description: as for outcome 38
Time Frame: Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 34 | 36 | 20 | 19
hours per day
  Month 6: Home healthcare services (n=0,2,0,0) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 2.00 (1.41) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point.
  Month 6: Work done (n=34,36,20,14) | 7.53 (2.19) | 10.36 (9.85) | 7.65 (2.16) | 10.21 (8.78)
  Month 6: Chores by housekeeper (n=8,9,9,5) | 2.88 (2.36) | 3.78 (1.20) | 5.00 (3.28) | 5.00 (1.58)
  Month 6: Chores by family/friend (n=31,22,18,19) | 3.16 (2.57) | 2.05 (1.05) | 2.72 (1.67) | 3.63 (5.58)
  Month 6: Missed work due to RA (n=3,3,0,3) | 4.00 (0.00) | 2.67 (1.15) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 2.00 (1.73)
  Month 6: RA related home HC services (n=0,2,0,0) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 1.00 (0.00) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point.

40. Secondary Outcome: Work Performance in Past 3 Months on Days Bothered as Assessed Using RA-HCRU at Baseline and Month 3
Description: Work performance of participants on number of days bothered was based on 10-point scale, where higher score indicated lower work performance.
Time Frame: Baseline, Month 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 73 | 76 | 73
units on a scale
  Baseline (n=73,76,72) | 4.27 (3.20) | 4.38 (3.12) | 4.65 (3.23)
  Month 3 (n=63,72,73) | 3.52 (3.24) | 3.51 (4.73) | 4.04 (3.37)

41. Secondary Outcome: Work Performance in Past 3 Months on Days Bothered as Assessed Using RA-HCRU at Month 6
Description: as for outcome 40
Time Frame: Month 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 59 | 63 | 33 | 29
units on a scale | 3.27 (2.94) | 2.63 (2.75) | 3.33 (3.22) | 4.83 (3.33)

42. Secondary Outcome: Work Limitations Questionnaire (WLQ) Score at Baseline and Month 3
Description: WLQ: participant-reported 25-item scale to evaluate degree to which health problems interfere with an ability to perform job roles along 4 dimensions: Time Management scale (TMS)(5-items); Physical Demands scale (PDS) (6-item); Mental-Interpersonal Demands Scale (MIDS) (9-items); Output Demands Scale (ODS) (5-items). All the scales ranged from 0 (limited none of the time) to 100 (limited all of the time). Work Loss Index (WLI), which represented percentage of lost work over time period relative to a normative population, was derived (total score: 0 [no loss] to 100 [complete loss of work]).
Time Frame: Baseline, Month 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 44 | 57 | 57
units on a scale
  Baseline: TMS (n=42,54,48) | 43.96 (26.39) | 48.53 (25.03) | 50.91 (28.08)
  Baseline: PDS (n=43,55,55) | 49.44 (28.49) | 48.95 (21.50) | 51.86 (25.25)
  Baseline: MIDS (n=42,54,56) | 28.44 (24.35) | 31.79 (23.66) | 34.36 (27.68)
  Baseline: ODS (n=41,50,52) | 41.95 (31.50) | 37.30 (25.74) | 40.20 (25.89)
  Baseline: WLI (n=44,57,57) | 10.51 (6.07) | 10.27 (5.71) | 10.99 (5.96)
  Month 3: TMS (n=38,50,42) | 36.09 (26.83) | 36.47 (26.72) | 47.62 (29.23)
  Month 3: PDS (n=40,51,43) | 52.08 (30.74) | 47.20 (26.39) | 42.31 (24.32)
  Month 3: MIDS (n=40,54,44) | 27.82 (28.80) | 28.60 (27.34) | 37.22 (28.70)
  Month 3: ODS (n=39,51,43) | 26.30 (29.16) | 30.78 (26.12) | 42.67 (28.97)
  Month 3: WLI (n=43,56,44) | 8.30 (6.57) | 8.73 (6.11) | 11.67 (6.29)

43. Secondary Outcome: Work Limitations Questionnaire (WLQ) Score at Month 6
Description: as for outcome 42
Time Frame: Month 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 40 | 45 | 24 | 19
units on a scale
  Month 6: TMS (n=39,42,23,18) | 26.96 (29.72) | 30.77 (27.83) | 32.50 (30.79) | 32.73 (25.10)
  Month 6: PDS (n=38,42,24,18) | 47.53 (36.97) | 44.65 (30.60) | 40.94 (27.82) | 47.15 (29.47)
  Month 6: MIDS (n=40,45,24,19) | 18.50 (26.90) | 29.84 (29.03) | 31.95 (32.26) | 30.68 (32.09)
  Month 6: ODS (n=39,44,24,19) | 21.32 (27.74) | 29.20 (29.00) | 30.50 (31.94) | 33.68 (28.02)
  Month 6: WLI (n=40,45,24,19) | 6.87 (6.53) | 8.78 (7.07) | 9.27 (7.06) | 9.62 (7.41)

44. Other Pre Specified Outcome: Number of Participants With Disease Activity Score Based on 28-Joints Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP]) Less Than 2.6 and Less Than or Equal to 3.2 at Week 2, Month 1 and 3
Description: DAS28-3 (CRP) was calculated from the SJC and TJC using the 28 joints count and CRP (mg/L). Total score range: 0-9.4, higher score=more disease activity. DAS28-3 (CRP) <=3.2 implied low disease activity and >3.2 to 5.1 implied moderate to high disease activity, and DAS28-3 (CRP) <2.6 = remission.
Time Frame: Week 2, Month 1, 3
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 132 | 133 | 131
participants
  Week 2: DAS28-3(CRP) <2.6 (n=127,125,124) | 8 | 12 | 2
  Week 2: DAS28-3(CRP) <=3.2 (n=127,125,124) | 19 | 23 | 4
  Month 1: DAS28-3(CRP) <2.6 (n=132,133,131) | 14 | 7 | 3
  Month 1: DAS28-3(CRP) <=3.2 (n=132,133,131) | 27 | 42 | 11
  Month 3: DAS28-3(CRP) <2.6 (n=132,133,131) | 27 | 35 | 6
  Month 3: DAS28-3(CRP) <=3.2 (n=132,133,131) | 45 | 57 | 13

45. Other Pre Specified Outcome: Number of Participants With Disease Activity Score Based on 28-Joints Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP]) Less Than 2.6 and Less Than or Equal to 3.2 at Month 4.5 and 6
Description: as for outcome 44
Time Frame: Month 4.5, 6
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 132 | 133 | 66 | 65
participants
  Month 4.5: DAS28-3(CRP) <2.6 | 31 | 42 | 14 | 12
  Month 4.5: DAS28-3(CRP) <=3.2 | 50 | 57 | 21 | 19
  Month 6: DAS28-3(CRP) <2.6 | 35 | 36 | 11 | 9
  Month 6: DAS28-3(CRP) <=3.2 | 57 | 59 | 23 | 19

46. Other Pre Specified Outcome: Number of Participants With Disease Activity Score Based on 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) Less Than 2.6 and Less Than or Equal to 3.2 at Month 3
Description: as for outcome 12
Time Frame: Month 3
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 119 | 125 | 120
participants
  Month 3: DAS28-4 (ESR) <2.6 | 8 | 14 | 2
  Month 3: DAS28-4 (ESR) <=3.2 | 17 | 28 | 6

47. Other Pre Specified Outcome: Number of Participants With Disease Activity Score Based on 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) Less Than 2.6 and Less Than or Equal to 3.2 at Month 6
Description: as for outcome 12
Time Frame: Month 6
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 122 | 127 | 63 | 60
participants
  Month 6: DAS28-4(ESR) <2.6 | 13 | 20 | 7 | 2
  Month 6: DAS28-4 (ESR) <=3.2 | 35 | 37 | 11 | 11

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- CP-690,550 5 mg Up to Month 3: CP-690,550 5 mg tablet orally twice daily up to Month 3.
- CP-690,550 10 mg Up to Month 3: CP-690,550 10 mg tablets orally twice daily up to Month 3.
- Placebo Up to Month 3: Placebo matching to CP-690,550 5 mg tablet orally twice daily up to Month 3.
- CP-690,550 5 mg From Month 3 to 6: CP-690,550 5 mg tablet orally twice daily from Month 3 to Month 6.
- CP-690,550 10 mg From Month 3 to 6: CP-690,550 10 mg tablets orally twice daily from Month 3 to Month 6.
Arm/Group | CP-690,550 5 mg Up to Month 3 | CP-690,550 10 mg Up to Month 3 | Placebo Up to Month 3 | CP-690,550 5 mg From Month 3 to 6 | CP-690,550 10 mg From Month 3 to 6
Serious Adverse Events (participants affected / at risk) | 2/133 | 2/134 | 6/132 | 8/199 | 8/200
Other Adverse Events (participants affected / at risk) | 37/133 | 43/134 | 46/132 | 35/199 | 30/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 5 mg Up to Month 3 (N=133) | CP-690,550 10 mg Up to Month 3 (N=134) | Placebo Up to Month 3 (N=132) | CP-690,550 5 mg From Month 3 to 6 (N=199) | CP-690,550 10 mg From Month 3 to 6 (N=200)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Ulcerative keratitis (Eye disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Drug ineffective (General disorders) | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Goodpasture's syndrome (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 5 mg Up to Month 3 (N=133) | CP-690,550 10 mg Up to Month 3 (N=134) | Placebo Up to Month 3 (N=132) | CP-690,550 5 mg From Month 3 to 6 (N=199) | CP-690,550 10 mg From Month 3 to 6 (N=200)
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 3 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 5 | 5 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 0
Nausea (Gastrointestinal disorders) | 4 | 2 | 9 | 4 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 6 | 3
Nasopharyngitis (Infections and infestations) | 5 | 6 | 4 | 6 | 5
Sinusitis (Infections and infestations) | 1 | 1 | 4 | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 5 | 2 | 4 | 5 | 8
Urinary tract infection (Infections and infestations) | 5 | 3 | 3 | 4 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 5 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 3 | 1 | 4 | 2
Fatigue (General disorders) | 1 | 3 | 0 | 0 | 0
Oedema peripheral (General disorders) | 3 | 1 | 5 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 3 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 5 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 2 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4 | 7 | 0
Headache (Nervous system disorders) | 3 | 8 | 1 | 1 | 4
Paraesthesia (Nervous system disorders) | 0 | 1 | 3 | 0 | 0
Depression (Psychiatric disorders) | 2 | 4 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.